CLINICAL TRIAL: NCT00856934
Title: A New Model to Enhance Wound Healing Using Autologous Keratinocytes in Platelet Concentrates - a Prospective Randomized Trial.
Brief Title: Effect of Platelet Rich Plasma and Keratinocyte Suspensions on Wound Healing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Wassim Raffoul / Medecin Chef, Service de Chirurgie Plastique et Reconstructrice, CHUV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132/03
Record Dates: First submitted 2009-01-02; First posted 2009-03-06 (Estimated); Results first posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-02

CONDITIONS: Skin Graft
Keywords: Skin graft donor site healing; skin; wound; platelet concentrate; keratinocytes; burns
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Wounds covered with standard dressings: three layers of paraffin gauze, standard bandages, elastic bandage.
  Interventions: Other: Standard dressings
- PRP (Experimental): PRP sprayed onto the wound bed with Calcium Choride. Wounds covered with same standard dressings used in control group.
  Interventions: Biological: Autologous Platelet Rich Plasma; Other: Standard dressings
- PRP+K (Experimental): Keratinocytes suspended in PRP sprayed onto the wound bed with Calcium Choride. Wounds covered with same standard dressings used in control group.
  Interventions: Biological: Autologous Platelet Rich Plasma; Biological: Keratinocyte suspension; Other: Standard dressings

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma — Platelet Rich Plasma isolated from patient blood sprayed onto wound bed along with 10% Calcium Chloride solution in a 10 to 1 proportion.
  Arms: PRP; PRP+K
Biological: Keratinocyte suspension — Autologous keratinocytes isolated from skin biopsy suspended in platelet rich plasma before spraying.
  Arms: PRP+K
Other: Standard dressings — Three layers of paraffin gauze, topped with standard dry bandages and an elastic bandage.

SUMMARY:
This prospective randomized trial evaluated the impact of autologous keratinocytes suspended in platelet concentrates on healing skin graft donor site wounds. It was hypothesized that the treatment would speed and improve wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Skin graft donor sites total surface < 15% BSA
* Skin graft donor site size: 0.2mm deep, 30 to 40 cm2 surface area

Exclusion Criteria:

* Patients treated with immunosuppressors
* Patients treated with corticoids
* Patients suffering from terminal renal insufficiency
* Patients suffering from severe peripheral arteriopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-06; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Raffoul, PD, MER, Principal Investigator — CHUV - CPR
Locations (1):
- Centre hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Fu X, Li X, Cheng B, Chen W, Sheng Z. Engineered growth factors and cutaneous wound healing: success and possible questions in the past 10 years. Wound Repair Regen. 2005 Mar-Apr;13(2):122-30. doi: 10.1111/j.1067-1927.2005.130202.x. PMID 15828936
- [Background] Ansel JC, Tiesman JP, Olerud JE, Krueger JG, Krane JF, Tara DC, Shipley GD, Gilbertson D, Usui ML, Hart CE. Human keratinocytes are a major source of cutaneous platelet-derived growth factor. J Clin Invest. 1993 Aug;92(2):671-8. doi: 10.1172/JCI116636. PMID 8349805
- [Background] Ballaun C, Weninger W, Uthman A, Weich H, Tschachler E. Human keratinocytes express the three major splice forms of vascular endothelial growth factor. J Invest Dermatol. 1995 Jan;104(1):7-10. doi: 10.1111/1523-1747.ep12613450. PMID 7798644
- [Background] Brown LF, Yeo KT, Berse B, Yeo TK, Senger DR, Dvorak HF, van de Water L. Expression of vascular permeability factor (vascular endothelial growth factor) by epidermal keratinocytes during wound healing. J Exp Med. 1992 Nov 1;176(5):1375-9. doi: 10.1084/jem.176.5.1375. PMID 1402682
- [Background] Decline F, Rousselle P. Keratinocyte migration requires alpha2beta1 integrin-mediated interaction with the laminin 5 gamma2 chain. J Cell Sci. 2001 Feb;114(Pt 4):811-23. doi: 10.1242/jcs.114.4.811. PMID 11171386
- [Background] Feliciani C, Gupta AK, Sauder DN. Keratinocytes and cytokine/growth factors. Crit Rev Oral Biol Med. 1996;7(4):300-18. doi: 10.1177/10454411960070040101. PMID 8986393
- [Background] McKay IA, Leigh IM. Epidermal cytokines and their roles in cutaneous wound healing. Br J Dermatol. 1991 Jun;124(6):513-8. doi: 10.1111/j.1365-2133.1991.tb04942.x. PMID 2064935
- [Background] Tamariz-Dominguez E, Castro-Munozledo F, Kuri-Harcuch W. Growth factors and extracellular matrix proteins during wound healing promoted with frozen cultured sheets of human epidermal keratinocytes. Cell Tissue Res. 2002 Jan;307(1):79-89. doi: 10.1007/s004410100450. Epub 2001 Nov 14. PMID 11810316
- [Background] Carter CA, Jolly DG, Worden CE Sr, Hendren DG, Kane CJ. Platelet-rich plasma gel promotes differentiation and regeneration during equine wound healing. Exp Mol Pathol. 2003 Jun;74(3):244-55. doi: 10.1016/s0014-4800(03)00017-0. PMID 12782011
- [Background] Knighton DR, Ciresi KF, Fiegel VD, Austin LL, Butler EL. Classification and treatment of chronic nonhealing wounds. Successful treatment with autologous platelet-derived wound healing factors (PDWHF). Ann Surg. 1986 Sep;204(3):322-30. doi: 10.1097/00000658-198609000-00011. PMID 3753059
- [Background] Mazzucco L, Medici D, Serra M, Panizza R, Rivara G, Orecchia S, Libener R, Cattana E, Levis A, Betta PG, Borzini P. The use of autologous platelet gel to treat difficult-to-heal wounds: a pilot study. Transfusion. 2004 Jul;44(7):1013-8. doi: 10.1111/j.1537-2995.2004.03366.x. PMID 15225241
- [Background] Valbonesi M, Giannini G, Migliori F, Dalla Costa R, Galli A. The role of autologous fibrin-platelet glue in plastic surgery: a preliminary report. Int J Artif Organs. 2002 Apr;25(4):334-8. doi: 10.1177/039139880202500413. PMID 12027145
- [Background] Brissett AE, Hom DB. The effects of tissue sealants, platelet gels, and growth factors on wound healing. Curr Opin Otolaryngol Head Neck Surg. 2003 Aug;11(4):245-50. doi: 10.1097/00020840-200308000-00005. PMID 14515071
- [Background] Feldman DL. Which dressing for split-thickness skin graft donor sites? Ann Plast Surg. 1991 Sep;27(3):288-91. doi: 10.1097/00000637-199109000-00017. PMID 1952757
- [Background] Gharaee-Kermani M, Phan SH. Role of cytokines and cytokine therapy in wound healing and fibrotic diseases. Curr Pharm Des. 2001 Jul;7(11):1083-103. doi: 10.2174/1381612013397573. PMID 11472255
- [Background] Werner S, Grose R. Regulation of wound healing by growth factors and cytokines. Physiol Rev. 2003 Jul;83(3):835-70. doi: 10.1152/physrev.2003.83.3.835. PMID 12843410
- [Background] Di Giulio AM, Picotti GB, Cesura AM, Panerai AE, Mantegazza P. Met-enkephalin immunoreactivity in blood platelets. Life Sci. 1982 May 10;30(19):1605-14. doi: 10.1016/0024-3205(82)90492-1. PMID 7098767
- [Background] Atiyeh BS, Gunn SW, Hayek SN. State of the art in burn treatment. World J Surg. 2005 Feb;29(2):131-48. doi: 10.1007/s00268-004-1082-2. PMID 15654666
- [Background] Hierner R, Degreef H, Vranckx JJ, Garmyn M, Massage P, van Brussel M. Skin grafting and wound healing-the "dermato-plastic team approach". Clin Dermatol. 2005 Jul-Aug;23(4):343-52. doi: 10.1016/j.clindermatol.2004.07.028. PMID 16023929
- [Background] Eaglstein WH, Falanga V. Chronic wounds. Surg Clin North Am. 1997 Jun;77(3):689-700. doi: 10.1016/s0039-6109(05)70575-2. PMID 9194887
- [Background] Edwards R, Harding KG. Bacteria and wound healing. Curr Opin Infect Dis. 2004 Apr;17(2):91-6. doi: 10.1097/00001432-200404000-00004. PMID 15021046
- [Background] Robson MC, Stenberg BD, Heggers JP. Wound healing alterations caused by infection. Clin Plast Surg. 1990 Jul;17(3):485-92. PMID 2199139
- [Background] Smith DJ Jr, Thomson PD, Garner WL, Rodriguez JL. Donor site repair. Am J Surg. 1994 Jan;167(1A):49S-51S. doi: 10.1016/0002-9610(94)90012-4. PMID 8109686
- [Result] Innes ME, Umraw N, Fish JS, Gomez M, Cartotto RC. The use of silver coated dressings on donor site wounds: a prospective, controlled matched pair study. Burns. 2001 Sep;27(6):621-7. doi: 10.1016/s0305-4179(01)00015-8. PMID 11525858
- [Result] Barnea Y, Amir A, Leshem D, Zaretski A, Weiss J, Shafir R, Gur E. Clinical comparative study of aquacel and paraffin gauze dressing for split-skin donor site treatment. Ann Plast Surg. 2004 Aug;53(2):132-6. doi: 10.1097/01.sap.0000112349.42549.b3. PMID 15269581
- [Result] Wiechula R. The use of moist wound-healing dressings in the management of split-thickness skin graft donor sites: a systematic review. Int J Nurs Pract. 2003 Apr;9(2):S9-17. doi: 10.1046/j.1322-7114.2003.00417.x. PMID 12694482
- [Result] Greenhalgh DG, Barthel PP, Warden GD. Comparison of back versus thigh donor sites in pediatric patients with burns. J Burn Care Rehabil. 1993 Jan-Feb;14(1):21-5. doi: 10.1097/00004630-199301000-00006. PMID 8454661
- [Result] Hart DW, Wolf SE, Herndon DN, Chinkes DL, Lal SO, Obeng MK, Beauford RB, Mlcak RT RP. Energy expenditure and caloric balance after burn: increased feeding leads to fat rather than lean mass accretion. Ann Surg. 2002 Jan;235(1):152-61. doi: 10.1097/00000658-200201000-00020. PMID 11753055
- [Result] Hormbrey E, Pandya A, Giele H. Adhesive retention dressings are more comfortable than alginate dressings on split-skin-graft donor sites. Br J Plast Surg. 2003 Jul;56(5):498-503. doi: 10.1016/s0007-1226(03)00195-4. PMID 12890465
- [Result] Rakel BA, Bermel MA, Abbott LI, Baumler SK, Burger MR, Dawson CJ, Heinle JA, Ocheltree IM. Split-thickness skin graft donor site care: a quantitative synthesis of the research. Appl Nurs Res. 1998 Nov;11(4):174-82. doi: 10.1016/s0897-1897(98)80296-6. PMID 9852660
- [Result] Bielecki TM, Gazdzik TS, Arendt J, Szczepanski T, Krol W, Wielkoszynski T. Antibacterial effect of autologous platelet gel enriched with growth factors and other active substances: an in vitro study. J Bone Joint Surg Br. 2007 Mar;89(3):417-20. doi: 10.1302/0301-620X.89B3.18491. PMID 17356164
- [Result] Moojen DJ, Everts PA, Schure RM, Overdevest EP, van Zundert A, Knape JT, Castelein RM, Creemers LB, Dhert WJ. Antimicrobial activity of platelet-leukocyte gel against Staphylococcus aureus. J Orthop Res. 2008 Mar;26(3):404-10. doi: 10.1002/jor.20519. PMID 17960651

RESULTS

PARTICIPANT FLOW:
Groups:
- PRP: Platelet Rich Plasma (PRP) sprayed onto the wound bed with Calcium Chloride. Wounds covered with same standard dressings used in control group.
- PRP+K: Keratinocytes suspended in Platelet Rich Plasma (PRP) sprayed onto the wound bed with Calcium Chloride. Wounds covered with same standard dressings used in control group.
Period: Overall Study
Arm/Group | Control | PRP | PRP+K
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PRP | PRP+K | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 12 | 41
  >=65 years | 0 | 1 | 3 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.9) | 45.5 (15.3) | 46.9 (20.5) | 44.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10 | 20
  Male | 11 | 9 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Complete Wound Healing
Description: Time required for complete epithelialization in days
Time Frame: Post operative day 5 and every other day thereafter
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control | PRP | PRP+K
Number analyzed (Participants) | 15 | 15 | 15
Days | 13.9 (2.0) | 7.2 (0.8) | 5.7 (0.7)
Statistical Analysis 1: Comparison: Control vs PRP vs PRP+K; Test type: Superiority or Other; p = 0.05, ANOVA

2. Secondary Outcome: Pain
Description: Pain evaluated on a Visual Analog Scale (VAS) from 0 (no pain) to 10 (extreme pain), specifically during dressing replacement.
Time Frame: Post operative day 5
Measure: Mean (Standard Deviation); unit: VAS Pain Score
Arm/Group | Control | PRP | PRP+K
Number analyzed (Participants) | 15 | 15 | 15
VAS Pain Score | 7.2 (0.7) | 1.5 (0.9) | 0.4 (0.7)
Statistical Analysis 1: Comparison: Control vs PRP vs PRP+K; Test type: Superiority or Other; p = 0.05, ANOVA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes